CLINICAL TRIAL: NCT01697358
Title: Prospective, Randomized Study of Multicolumn Implantable Lead Stimulation for Predominant Low Back Pain
Brief Title: Spinal Cord Stimulation for Predominant Low Back Pain
Acronym: PROMISE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1665
Record Dates: First submitted 2012-09-25; First posted 2012-10-02 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-06

CONDITIONS: Failed Back Surgery Syndrome; Back Pain; Pain in Leg, Unspecified
Keywords: FBSS; post laminectomy syndrome; SCS; RCT; back pain
MeSH Terms: conditions — Failed Back Surgery Syndrome; Back Pain; post laminectomy syndrome | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Intervention Model Description: Period I (from randomization to 6 months) is the randomized parallel group comparative phase. Day zero for the study is the point of randomization. The randomization ratio is 1:1 (SCS+OMM to OMM). For the SCS+OMM arm, the screening test and/or implant occurred after randomization. Period II (6 to 24 months) is the long-term observational follow-up phase.
Oversight: Data Monitoring Committee: No

ARMS (2):
- SCS + OMM (Active Comparator): Spinal Cord Stimulation (SCS) using the Medtronic Specify 5-6-5 multicolumn surgical lead plus an individual Optimal Medical Management (OMM) treatment plan
  Interventions: Device: Spinal Cord Stimulation (SCS); Drug: Optimal Medical Management (OMM)
- OMM alone (Active Comparator): The investigator and subject will determine an individual Optimal Medical Management (OMM) treatment plan
  Interventions: Drug: Optimal Medical Management (OMM)

INTERVENTIONS:
Device: Spinal Cord Stimulation (SCS) — Spinal Cord Stimulation (SCS) using the Medtronic Specify 5-6-5 multicolumn surgical lead. Subjects will undergo an SCS screening test and, if successful, an implantable neurostimulation system implant. Any SCS group subject not implanted will continue to be treated with OMM and will be followed as part of the SCS group.
  Arms: SCS + OMM
Drug: Optimal Medical Management (OMM) — The investigator and subject will determine an individual OMM treatment plan, which should include non-investigational pharmacologic agents and/or therapies.

SUMMARY:
The purpose of this study is to compare the effectiveness of spinal cord stimulation (SCS) using the Medtronic Specify® 5-6-5 multicolumn surgical lead plus optimal medical management (OMM) versus OMM alone in patients suffering from predominant low back pain due to failed back surgery syndrome (FBSS).

DETAILED DESCRIPTION:
The study has a multi-center, prospective, randomized (1:1), open-label, parallel-group design of two alternative treatments:

* SCS group (SCS+OMM)
* OMM group

ELIGIBILITY:
Inclusion Criteria:

* SCS candidate with the Specify 5-6-5 surgical lead
* Has FBSS and does not require further surgery (defined as persistent or recurrent low back and leg pain of at least 6 months duration following at least one decompression and/or fusion procedure)
* Average low back pain is ≥ 5 as assessed by the baseline NPRS
* Average low back pain is greater than leg pain
* Subject has persistent moderate to severe low back and leg pain despite other treatments

Exclusion Criteria:

* Treated with SCS, subcutaneous or peripheral nerve stimulation, an intrathecal drug delivery system, requires back surgery at the location related to his/her original back pain complaint or experimental therapies
* Most recent back surgery < 6 months ago
* Low back pain only (no leg pain)
* Investigator suspects substance abuse that might confound the study results
* Radiographic evidence of instability requiring fusion
* Pain relieved completely by lying down
* Life expectancy of < 24 months
* Subject is pregnant or planning to become pregnant during the course of the study
* Subject is unable to undergo study assessments or complete questionnaires independently

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2013-01-08 (Actual); Primary Completion 2016-03-12 (Actual); Study Completion 2017-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Rigoard, MD, PhD, Study Chair — University of Poitiers
Locations (28):
- United States (12):
  - Pain Care LLC, Stockbridge, Georgia
  - The Neuroscience Center, Ocean Springs, Mississippi
  - Kozmary Center for Pain Management, Las Vegas, Nevada
  - Albany Medical College, Albany, New York
  - Weill Medical College of Cornell University, New York, New York
  - New York Spine and Wellness Center, North Syracuse, New York
  - University of Rochester Neurosurgery Partners in Pain Management, Rochester, New York
  - Duke Spine Center, Durham, North Carolina
  - WellSpan Interventional Pain Center, York, Pennsylvania
  - Richmond Bone and Joint Clinic, Sugar Land, Texas
  - Utah Spine Care, Ogden, Utah
  - West Virginia University, Morgantown, West Virginia
- Belgium (5):
  - UCL St. Luc, Brussels
  - AZ St. Maarten, Duffel
  - CHR Citadelle, Liège
  - Heilig Hart Ziekenhuis, Roeselare
  - Department of Neurosurgery: St. Augustinus Ziekenhuizen, Wilrijk
- Regina General Hospital, Regina, Canada
- Colombia (3):
  - Clínica Las Américas, Medellín, Antioquia
  - Hospital Pablo Tobón Uribe, Medellín, Antioquia
  - San Vicente Fundación, Rionegro, Antioquia
- Centre Hospitalier Universitaire de Poitiers, Poitiers, France
- Städtisches Klinikum Görlitz gGmbH, Görlitz, Germany
- St. Elisabeth Ziekenhuis Tilburg, Tilburg, Netherlands
- Spain (2):
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
- United Kingdom (2):
  - Nottingham University Hospital NHS Trust, Nottingham
  - John Radcliffe Hospital Oxford, Oxford

IPD SHARING:
Plan to Share IPD: No
Data will be kept confidential by Medtronic and only be shared with study investigators following Medtronic approval of a data request form.

REFERENCES:
- [Derived] O'Connell NE, Ferraro MC, Gibson W, Rice AS, Vase L, Coyle D, Eccleston C. Implanted spinal neuromodulation interventions for chronic pain in adults. Cochrane Database Syst Rev. 2021 Dec 2;12(12):CD013756. doi: 10.1002/14651858.CD013756.pub2. PMID 34854473
- [Derived] Rigoard P, Basu S, Desai M, Taylor R, Annemans L, Tan Y, Johnson MJ, Van den Abeele C, North R; PROMISE Study Group. Multicolumn spinal cord stimulation for predominant back pain in failed back surgery syndrome patients: a multicenter randomized controlled trial. Pain. 2019 Jun;160(6):1410-1420. doi: 10.1097/j.pain.0000000000001510. PMID 30720582
- [Derived] Rigoard P, Desai MJ, North RB, Taylor RS, Annemans L, Greening C, Tan Y, Van den Abeele C, Shipley J, Kumar K. Spinal cord stimulation for predominant low back pain in failed back surgery syndrome: study protocol for an international multicenter randomized controlled trial (PROMISE study). Trials. 2013 Nov 7;14:376. doi: 10.1186/1745-6215-14-376. PMID 24195916

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 278 subjects were recruited between January 2013 and August 2015 from 28 sites in Canada, Colombia, Europe, and US.
Pre-assignment Details: A total of 60 subjects didn't meet the inclusion and/or exclusion criteria and discontinued from the study before randomization.
Groups:
- SCS + OMM: Spinal Cord Stimulation (SCS) using multicolumn surgical lead + Optimal Medical Management (OMM): In addition to the OMM described under the OMM group, subjects underwent an SCS screening test and, if successful, received an INS implant. Any SCS group subject not implanted continued to be treated with OMM and were followed as part of the SCS group.
- OMM Alone: Optimal Medical Management (OMM) alone: Pain treatment was evaluated, and medical management of subjects' pain was optimized. The investigator and subject determined an individual OMM treatment plan, which should include non-investigational pharmacologic agents (e.g., tricyclic antidepressants, opioid analgesics or tramadol, antiepileptics, or lidocaine) and/or interventional therapies (e.g., therapeutic injections, radiofrequency, acupuncture, and physical therapy) as appropriate. Excluded from OMM is intrathecal drug delivery (IDD), peripheral nerve stimulation (PNS; not an approved indication in the USA), back surgery at the location related to the subject's original back pain complaint and experimental therapies. Data regarding pain treatments implemented during the study were collected to reveal how medical management was optimized.
Period: Period I: Randomization to 6 Months
Arm/Group | SCS + OMM | OMM Alone
Started | 110 | 108
Completed | 97 | 107
Not Completed | 13 | 1
Not completed — Withdrawal by Subject | 6 | 0
Not completed — Physician Decision | 4 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 2 | 0
Period: Period II: 6-24M Long-term Follow-up
Arm/Group | SCS + OMM | OMM Alone
Started | 97 | 107
Completed | 48 | 52
Not Completed | 49 | 55
Not completed — Physician Decision | 3 | 12
Not completed — Withdrawal by Subject | 8 | 10
Not completed — Lost to Follow-up | 3 | 3
Not completed — Death | 1 | 1
Not completed — Adverse Event | 0 | 3
Not completed — Active subjects at the time of posting | 34 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SCS + OMM | OMM Alone | Total
Number analyzed (Participants) | 110 | 108 | 218
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.8 (12.5) | 55.1 (10.2) | 53.9 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 64 | 132
  Male | 42 | 44 | 86
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 25 | 24 | 49
  Canada | 4 | 4 | 8
  Colombia | 6 | 4 | 10
  France | 12 | 13 | 25
  Germany | 2 | 2 | 4
  Netherlands | 6 | 6 | 12
  Spain | 5 | 6 | 11
  United Kingdom | 18 | 17 | 35
  United States | 32 | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: Compare Proportion of Subjects With ≥50% Reduction in Low Back Pain Intensity Between the Treatment Groups
Description: Compare the proportion of subjects with a ≥50% reduction in low back pain intensity, as measured by the NPRS, from baseline to the end of Period I in the SCS group with that in the OMM group. Subjects reported average low back pain using a 11-point NPRS pain diary (0 = no back pain, 10 = worst low back pain imaginable) two times per day for a 7-day period at baseline and prior to 6-month visit. Percent reduction in low back pain intensity was calculated as average NPRS at (6-month visit - baseline) / baseline. Subjects with ≥50% reduction in average low back pain were considered as responders.
Time Frame: 6 months post randomization
Population: Intent-to-treat (ITT) - included all randomized subjects and analyzed as randomized, regardless the subjects' status at 6 months. Subjects in the SCS+OMM group received screening tests after the randomization, and might not have proceeded to implant of the neurostimulator. Subjects with missing data at 6 months were imputed as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | SCS + OMM | OMM Alone
Number analyzed (Participants) | 110 | 108
Participants | 15 | 5
Statistical Analysis 1: Comparison: SCS + OMM vs OMM Alone; Test type: Superiority; p = 0.036, Z-test using unpooled standard deviation

2. Secondary Outcome: Compare Change in Low Back Pain Intensity, as Measured by the Numeric Pain Rating Scale (NPRS), Between the Treatment Groups
Description: Compare change in low back pain intensity, as measured by the Numeric Pain Rating Scale (NPRS), from baseline to the end of Period I for subjects in the SCS group with that in the OMM group. Subjects reported average low back pain using a 11-point NPRS pain diary (0 = no back pain, 10 = worst low back pain imaginable) two times per day for a 7-day period at baseline and prior to 6-month visit. Change in low back pain intensity is calculated as NPRS at baseline - NPRS at 6-month visit, with a positive change indicated as an improvement.
Time Frame: 6 months post randomization
Population: Intent-to-treat (ITT) - included all randomized subjects and analyzed as randomized, regardless the subjects' status at 6 months. Subjects in the SCS+OMM group received screening tests after the randomization, and might not have proceeded to implant of the neurostimulator. Subjects with missing data at 6 months were imputed as having no change.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SCS + OMM | OMM Alone
Number analyzed (Participants) | 110 | 108
units on a scale | 1.4 (1.9) | 0.3 (1.7)
Statistical Analysis 1: Comparison: SCS + OMM vs OMM Alone; Test type: Superiority; p < 0.001, Regression, Linear; Variables included in the linear regression model are: baseline NPRS, treatment group, and virtual center

3. Secondary Outcome: Compare Change in Leg Pain Intensity, as Measured by the NPRS, Between the Treatment Groups
Description: Compare change in leg pain intensity, as measured by the NPRS, from baseline to the end of Period I for subjects in the SCS group with that in the OMM group. Subjects reported average leg pain using a 11-point NPRS pain diary (0 = no back pain, 10 = worst low back pain imaginable) two times per day for a 7-day period at baseline and prior to 6-month visit. Change in leg pain intensity is calculated as NPRS at baseline - NPRS at 6-month visit, with a positive change indicated as an improvement.
Time Frame: 6 months post randomization
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SCS + OMM | OMM Alone
Number analyzed (Participants) | 110 | 108
units on a scale | 1.2 (2.1) | -0.1 (2.4)
Statistical Analysis 1: Comparison: SCS + OMM vs OMM Alone; Test type: Superiority; p < 0.001, Regression, Linear; Variables included in the linear regression model are: baseline NPRS, treatment group, and virtual center

4. Secondary Outcome: Compare Change in Functional Disability, as Measured by the Oswestry Disability Index (ODI), Between the Treatment Groups
Description: ODI is a validated questionnaire of 10 subject-reported sections on the ability to perform activities of daily living. These 10 sections are pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life (if applicable), social life, and traveling. Each section was scored on a 0 to 5 scale with 0 indicating no limitation of function due to pain and 5 indicating major functional disability due to back pain. A raw ODI score was calculated from the total score of 10 sections (minimum is 0 and maximum is 50). This ODI raw score was then normalized to a scale of 0 to 100, with 0-20 categorized as minimal disability, 20-40 as moderate disability, 40-60 as severe disability, 60-80 as severely disabled, and 80-100 as bed-bound patients. The ODI was assessed at baseline and subsequent scheduled study visits. Change in functional disability is calculated as ODI at baseline - ODI at 6-month visit, with a positive change indicated as an improvement.
Time Frame: 6 months post randomization
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SCS + OMM | OMM Alone
Number analyzed (Participants) | 110 | 108
units on a scale | 8.1 (14.7) | 1.8 (14.3)
Statistical Analysis 1: Comparison: SCS + OMM vs OMM Alone; Test type: Superiority; p < 0.001, Regression, Linear; Variables included in the linear regression model are: baseline ODI, treatment group, and virtual center

5. Secondary Outcome: Compare Change in Quality of Life (QoL), as Measured by the SF-36 Physical Component Summary (PCS), Between the Treatment Groups
Description: The QoL scores were collected using the SF-36 questionnaire, which included the scores in the following 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, mental health. The raw score of 0 represents poor health and 100 represents best health. The Physical Component Summary (PCS) score is a norm based score calculated from the raw scores of these 8 domains with a focus on physical health using 1998 US population. Change in PCS is calculated as PCS at 6-month visit - PCS at baseline, with a positive change indicated as an improvement.
Time Frame: 6 months post randomization
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SCS + OMM | OMM Alone
Number analyzed (Participants) | 110 | 108
units on a scale | 5.27 (8.28) | 1.34 (6.28)
Statistical Analysis 1: Comparison: SCS + OMM vs OMM Alone; Test type: Superiority; p < 0.001, Regression, Linear; Variables included in the linear regression model are: baseline PCS, treatment group, and virtual center

6. Other Pre Specified Outcome: Compare Proportion of Subjects With ≥30% Reduction in Low Back Pain Intensity Between the Treatment Groups
Description: This additional analysis was pre-specified to support the analysis of primary objective. The 30% responder which is defined in the following paragraph was considered as clinical relevant to the SCS therapy in back pain. Compare the proportion of subjects with a ≥30% reduction in low back pain intensity, as measured by the NPRS, from baseline to the end of Period I in the SCS group with that in the OMM group. Subjects reported average low back pain using a 11-point NPRS pain diary (0 = no back pain, 10 = worst low back pain imaginable) two times per day for a 7-day period at baseline and prior to 6-month visit. Percent reduction in low back pain intensity was calculated as average NPRS at (6-month visit - baseline) / baseline. Subjects with ≥30% reduction in average low back pain were considered as 30% responders.
Time Frame: 6 months post randomization
Population: As-treated - included all randomized subjects who provided data at 6-month visit, and analyzed based on the actual treatment the subjects received at 6-month visit.
Measure: Count of Participants; unit: Participants
Arm/Group | SCS + OMM | OMM Alone
Number analyzed (Participants) | 79 | 117
Participants | 31 | 14
Statistical Analysis 1: Comparison: SCS + OMM vs OMM Alone; Test type: Superiority; p < 0.001, Z-test using unpooled standard deviation

ADVERSE EVENTS:
Time Frame: Randomization to 6 months
Arm/Group | SCS + OMM | OMM Alone
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/108
Serious Adverse Events (participants affected / at risk) | 18/110 | 7/108
Other Adverse Events (participants affected / at risk) | 4/110 | 11/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCS + OMM (N=110) | OMM Alone (N=108)
Implant site infection (Infections and infestations) | 6 (7) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Drug abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Implant site pain (General disorders) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Device extrusion (Product Issues) | 0 (0) | 1 (1)
Device stimulation issue (Product Issues) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCS + OMM (N=110) | OMM Alone (N=108)
Adverse drug reaction (General disorders) | 2 (2) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No